CLINICAL TRIAL: NCT05296265
Title: Efficacy and Mechanisms of Virtual Reality Treatment of Phantom Leg Pain: In-Person Treatment
Brief Title: Efficacy and Mechanisms of Virtual Reality Treatment of Phantom Leg Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: University of Pennsylvania (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Laurel Buxbaum, Associate Director, Moss Rehabilitation Research Institute, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-775.
Record Dates: First submitted 2022-02-09; First posted 2022-03-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-05

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: Forty individuals with above (AKA) or below (BKA) knee amputation suffering from chronic phantom limb pain (PLP) will be recruited and will be quasi-randomly assigned to Active VR versus Distractor VR treatments in 50:50 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active VR treatment (Experimental): Subjects assigned to the Active VR treatment will begin by selecting an avatar, with features such as gender and skin color that can be chosen according to preference. During treatment, they will participate in a variety of games and activities developed and used by our teams including Kick, Dog Food, Quest for Fire, Chess, Checkers, Sudoku, and surfing the internet. Subjects will have substantial flexibility to select games according to their interests but will be required to spend at least 30 minutes in each session in games that require forceful, large amplitude, movements of the amputated lower limb (e.g., Quest for Fire, Kick). Time spent and level of engagement as measured by movements of the avatar or, in the case of chess, checkers, solitaire, Sudoku, and internet surfing, the number of clicks produced with each leg will be recorded for each activity using custom software
  Interventions: Behavioral: VR treatment for phantom limb pain
- Distractor VR treatment (Experimental): Subjects assigned to the Distractor VR treatment will participate in REAL i-Series immersive VR experience (REAL system), which has been demonstrated to reduce pain in several studies but lacks the hypothesized "active ingredients" of our Active VR treatment (visual and auditory feedback of movement of an extrapolated amputated limb). Subjects will navigate through pleasant and relaxing VR environments; they will not see any rendering of their body and make no movements with their legs
  Interventions: Behavioral: VR treatment for phantom limb pain

INTERVENTIONS:
Behavioral: VR treatment for phantom limb pain — 8 twice-weekly interventions of 1 hour; baseline, pre-intervention; immediately after the end of the in intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention

SUMMARY:
After amputation of an arm or leg, up to 90% of subjects experience a "phantom limb", a phenomenon characterized by persistent feelings of the missing limb. Many subjects with a phantom limb experience intense pain in the missing extremity that is often poorly responsive to medications or other interventions. The proposed work will contrast the efficacy of two virtual reality treatments for phantom limb pain: a 'Distractor' and an Active VR treatment. In the Distractor treatment, participants are engaged in a visually immersive virtual reality experience that does not require leg movements (REAL i-Series® immersive VR experience). In the Active VR treatment, subjects play a series of VR games using the virtual rendering of both legs.

DETAILED DESCRIPTION:
Almost 2 million people in the US have had an amputation and up to 90% of people with limb amputation experience the persistent sensation of the missing extremity, a phenomenon known as a "phantom limb" (Weeks et al., 2010). Additionally, a significant proportion of individuals with a phantom limb - up to 85% in some studies - experience persistent and debilitating pain in the missing limb, a condition known as phantom limb pain (hereafter PLP). Although existing therapies provide pain relief in some cases, there is widespread agreement that current approaches fall short of bringing relief to most individuals with PLP (Weeks et al., 2010).

The investigators recently completed a proof-of-concept study (Ambron et al., 2021) in which eight subjects with below knee amputations (BKA) underwent two virtual reality (VR) treatments for PLP. In an Active VR treatment, subjects played a variety of active games requiring leg movements while receiving high-quality visual feedback of the missing lower leg. Feedback about leg position was provided via an electromagnetic system using leg sensors (trackSTAR, Ascension Technologies Inc), and the program generated an image of the missing lower leg, visible as a first-person avatar. This treatment was contrasted with a "Distractor" treatment, in which participants were engaged in a visually immersive virtual reality experience that did not require leg movements (Cool!TM). Both treatments were associated with significant reductions in pain intensity, but the Active VR treatment was also associated with reductions in pain interference, depression, and anxiety.

The specific aims of the current study are (i) to replicate our prior observations of efficacy of VR treatment in a larger sample of individuals with BKA; (ii) to test VR therapy in patients with above knee amputations; (iii) to compare the efficacy of Active VR treatment to Distractor VR treatment for PLP on measures of pain as well as psychological health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 100 years
2. Capacity to provide Informed Consent
3. Unilateral above or below knee amputation more than 3 months prior to enrollment
4. Absence of cognitive impairment, operationally defined as a Montreal Cognitive Assessment score of 18 or greater
5. Pain averaged over the preceding 1 month in the phantom limb rated as greater than 4 on a scale of 0-10.

Exclusion Criteria:

1. History of significant medical or neurological disorder such as stroke or moderate to severe traumatic brain injury (operationally defined as loss of consciousness for more than 30 minutes)
2. History of significant or poorly controlled psychiatric disorders
3. Current significant depression or anxiety as judged by the Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983).
4. Current abuse of alcohol or drugs, prescription or otherwise
5. Nursing a child, pregnant, or intent to become pregnant during the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | pre each intervention (8 sessions); immediately after each intervention (8 session); baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  Visual Analogue Scale of McGill Short Form Questionnaire (Melzack, 1987); 0 minimum score - 10 maximum score; higher scores indicate higher level of pain (worse outcome)
Changes in pain quality | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  McGill Short Form Questionnaire (Melzack, 1987): a series of 4-point scales assessing 15 characteristics of pain (e.g., throbbing, shooting, cramping, etc.). It generates separate scores for Sensory, Affective, and Total pain (maximum 78 points), and correlates strongly with the well-known long form of the questionnaire

SECONDARY OUTCOMES:
Changes in average pain after the treatment | up to 4 weeks
  average pain intensity since the previous intervention on an 11-point numerical rating pain scale; (0 - minimum score/no pain; 10 maximum score/pain as bad as participants can imagine); higher scores indicate higher level of pain (worse outcome)

OTHER OUTCOMES:
Changes in daily activities after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Frenchay Activities Index (FAI) (Holbrook et al., 1983):1983): a scale measuring the physical function and daily activity that has excellent reliability in subjects with lower-limb amputation in predicting quality of life (Asono et al., 2008). 0 minimum score - 45 maximum score; higher scores indicate more daily activities (better outcome).
Changes in quality of life after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The 12-Item Short Form Health Survey (SF-12) (Ware et al., 1996): a brief measure of quality of life and functional capacity that has been validated in patients with amputation and PLP (Padovani et al., 2015; Chen et al., 2012; Pape et al., 2010). 0 minimum score - 100 maximum score. Higher scores indicate lower physical and mental health (worse outcome).
Changes in pain interference after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Pain Interference Scale from the Brief Pain Inventory (BPI) (Cleeland & Ryan, 1994): this assesses the degree to which pain interferes with daily activities using a 0-10 numeric rating scale. 0 minimum score - 10 maximum score. Higher scores indicate higher pain interference (worse outcome).
Changes in depression and anxiety as effect of the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983):1983): the HADS is a 14- item measure assessing both depressive and anxiety symptoms. In addition to providing separate scores for anxiety and depression, the HADS also provides a measure of global negative affect. 0 minimum score - 42 maximum score. Higher scores indicate more depression and anxiety (worse outcome)
Changes in the pain catastrophizing after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The 13-item Pain Catastrophizing Scale (Sullivan et al., 1995): this scale investigates pain catastrophizing, which has been highly associated with pain severity and disability after amputation (Hanley et al., 2004; Whyte & Carroll, 2004; Jensen et al., 2002). 0 minimum score -52; Higher scores indicate higher tendency to catastrophizing (worse outcome)
Changes in insomnia after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  Insomnia Severity Index (Bastien et al., 2001): this is a 7-point scale that measure insomnia, a symptom associated with PLP (Durmus et al., 2015). 0 minimum score - 28 maximum score; higher scores indicate more insomnia (worse outcome)
Perception of VR system | baseline, pre-intervention
  Technology Acceptance Scale (Morris et al., 1997): this is a 7-point scale that measure level of acceptance of the VR system. 0 minimum score - 133 maximum score; higher scores indicate low level of acceptance (worse score)
Usability of each game | immediately after the last intervention (session 8 of the intervention);
  System Usability Scale (SUS) (Brooke, 1996); Scale measuring the usability of each game; minimum score 10 - maximum score 50. Higher scores indicate less usability (worse outcome).
Cybersickness | day 1, day 8
  Simulator Sickness Questionnaire (Kennedy et al., 1993);
Presence in VR | day 1, day 8
  Brief Slater-Usoh-Steed Presence Questionnaire (Usoh et al., 2000; Slater et al., 1998; 1994). 7 minimum score - 42 maximum score. Higher scores indicate more presence in the VR (better outcome
Changes in PL and PLP after the treatment | baseline, pre-intervention; immediately after the end of the intervention; 1 week after the end of the intervention; 8 weeks after the end of the intervention
  The Modified Limb Deficiency and Phantom Limb Questionnaire (Goller et al., 2013): this questionnaire assesses prosthesis type and usage and non-painful phantom limb experiences, including perceived position (e.g., telescoping) and ability to move the phantom. In addition to providing useful descriptive information, prosthesis use and telescoping will be used in the adaptive randomization algorithm to assign subjects to treatments.
Treatment satisfaction | 1 week after the end of the intervention
  visual analogue scale that evaluates treatment satisfaction (Robinson et al., 2004; Smith et al., 2005); 0 minimum score - 10 maximum score; Higher scores indicate more treatment satisfaction (better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Buxbaum, PsyD, Principal Investigator — Albert Einstein Healthcare Netork
Locations (3):
- United States (3):
  - Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington-Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
After de-identification, individual participant data to be shared will include descriptors of clinical status (e.g., time since amputation, level of amputation), background test battery results, and outcome measures results.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a sound rationale.

REFERENCES:
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Holbrook M, Skilbeck CE. An activities index for use with stroke patients. Age Ageing. 1983 May;12(2):166-70. doi: 10.1093/ageing/12.2.166. PMID 6869117
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Goller AI, Richards K, Novak S, Ward J. Mirror-touch synaesthesia in the phantom limbs of amputees. Cortex. 2013 Jan;49(1):243-51. doi: 10.1016/j.cortex.2011.05.002. Epub 2011 Jun 22. PMID 22981809
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Slater M, Steed A, McCarthy J, Maringelli F. The influence of body movement on subjective presence in virtual environments. Hum Factors. 1998 Sep;40(3):469-77. doi: 10.1518/001872098779591368. PMID 9849105
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Ambron E, Buxbaum LJ, Miller A, Stoll H, Kuchenbecker KJ, Coslett HB. Virtual Reality Treatment Displaying the Missing Leg Improves Phantom Limb Pain: A Small Clinical Trial. Neurorehabil Neural Repair. 2021 Dec;35(12):1100-1111. doi: 10.1177/15459683211054164. Epub 2021 Oct 27. PMID 34704486
- [Background] Robinson LR, Czerniecki JM, Ehde DM, Edwards WT, Judish DA, Goldberg ML, Campbell KM, Smith DG, Jensen MP. Trial of amitriptyline for relief of pain in amputees: results of a randomized controlled study. Arch Phys Med Rehabil. 2004 Jan;85(1):1-6. doi: 10.1016/s0003-9993(03)00476-3. PMID 14970960
- [Background] Smith DG, Ehde DM, Hanley MA, Campbell KM, Jensen MP, Hoffman AJ, Awan AB, Czerniecki JM, Robinson LR. Efficacy of gabapentin in treating chronic phantom limb and residual limb pain. J Rehabil Res Dev. 2005 Sep-Oct;42(5):645-54. doi: 10.1682/jrrd.2005.05.0082. PMID 16586190